CLINICAL TRIAL: NCT03506698
Title: Kangaroo Mother Care Implementation Research for Accelerating Scale-up
Status: Completed | Type: Observational
Sponsor: Rajiv Bahl (Other)
Collaborators: Mekelle University (Other); Emory University (Other); Emory University Ethiopia (Unknown); Hawassa University (Other)
Responsible Party: Sponsor-Investigator, Rajiv Bahl, Study Director, World Health Organization
Organization: World Health Organization (Other)
Other Study IDs: ERC.0002716
Record Dates: First submitted 2018-03-22; First posted 2018-04-24 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Low Birth Weight
Keywords: Birth weight
MeSH Terms: conditions — Birth Weight | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Kangaroo Mother Care (KMC) — Skin to skin contact of newborns with mothers or caregiver for a minimum of at least eight hours over a 24-hours period, along with exclusive breastfeeding or breast milk feeding via tube or spoon

SUMMARY:
The implementation research project aims to develop and evaluate models for scaling up KMC in health facilities across India and Ethiopia and thereby develop effective approaches to achieve high population coverage

DETAILED DESCRIPTION:
Kangaroo Mother Care (KMC) is the practice of early, continuous and prolonged skin-to-skin contact between the mother and the baby with exclusive breastfeeding. Despite clear evidence of impact in improving survival and health outcomes among low birth weight infants, KMC coverage has remained low and implementation has been limited. The multi-site project includes formative research to identify barriers and contextual factors that affect implementation and utilization of KMC and design scalable models to deliver KMC across the facility-community continuum. This will be followed by implementation and evaluation of these models in routine care settings, in an iterative fashion, with the aim of reaching a successful model for wider district, state and national-level scale-up. The aim is to successfully provide KMC to 80% or more of babies born in the study area weighing under 2000 grammes

ELIGIBILITY:
Inclusion Criteria:

• All newborns who are less than 2000 gm born within the study facilities during the study period.

Exclusion Criteria:

• Newborns who are sick per predefined criteria will not be provided KMC until they have been stabilized. Criteria for delay of initiation include: critical illness including apnea, decreased respiratory rate <20 breaths per minute, grunting, cyanosis, severe chest in-drawing, convulsions, unconsciousness, and severe hypothermia <32°F.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborn babies with birth weight less than 2000gm born in the geographic area targeted by the intervention, including all babies born in health facilities and in the community
Sampling Method: Non-Probability Sample
Enrollment: 3804 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Effective coverage of KMC at 7 days after discharge | 7 days after discharge
  Effective coverage will be defined as adoption of skin-to-skin care for at least 8 hours and exclusive breastfeeding in the 24 hours prior to assessment

CONTACTS AND LOCATIONS:
Overall Officials: Araya Abrha Medhanyie, PhD, Principal Investigator — Mekelle University; Abebe Gebremariam Gobezayehu, MD, Principal Investigator — Emory University Ethiopia; John Cranmer, DNP, MPH, Principal Investigator — Emory University; Henok Tadele Dangiso, MD, Principal Investigator — Hawassa University
Locations (3):
- Ethiopia (3):
  - Hawassa University Referral Hospital, Awasa
  - Felege Hiwot Hospital, Bahir Dar
  - Ayder Comprehensive Specialized Hospital, Mek'ele

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mony PK, Tadele H, Gobezayehu AG, Chan GJ, Kumar A, Mazumder S, Beyene SA, Jayanna K, Kassa DH, Mohammed HA, Estifanos AS, Kumar P, Jadaun AS, Hailu Abay T, Washington M, W/Gebriel F, Alamineh L, Fikre A, Kumar A, Trikha S, Ashebir Gebregizabher F, Kar A, Bilal SM, Belew ML, Debere MK, Krishna R, Dalpath SK, Amare SY, Mohan HL, Brune T, Sibley LM, Tariku A, Sahu A, Kumar T, Hadush MY, Gowda PD, Aziz K, Duguma D, Singh PK, Darmstadt GL, Agarwal R, Gebremariam DS, Martines J, Portela A, Jaiswal HV, Bahl R, Rao Pn S, Tadesse BT, Cranmer JN, Hailemariam D, Kumar V, Bhandari N, Medhanyie AA; KMC Scale-Up Study Group. Scaling up Kangaroo Mother Care in Ethiopia and India: a multi-site implementation research study. BMJ Glob Health. 2021 Sep;6(9):e005905. doi: 10.1136/bmjgh-2021-005905. PMID 34518203
- [Derived] Medhanyie AA, Alemu H, Asefa A, Beyene SA, Gebregizabher FA, Aziz K, Bhandari N, Beyene H, Brune T, Chan G, Cranmer JN, Darmstadt G, Duguma D, Fikre A, Andualem BG, Gobezayehu AG, Mariam DH, Abay TH, Mohan HL, Jadaun A, Jayanna K, Kajal FNU, Kar A, Krishna R, Kumar A, Kumar V, Madhur TK, Belew ML, M R, Martines J, Mazumder S, Amin H, Mony PK, Muleta M, Pileggi-Castro C, Pn Rao S, Estifanos AS, Sibley LM, Singhal N, Tadele H, Tariku A, Lemango ET, Tadesse BT, Upadhyay R, Worku B, Hadush MY, Bahl R; KMC Scale-Up Study Group. Kangaroo Mother Care implementation research to develop models for accelerating scale-up in India and Ethiopia: study protocol for an adequacy evaluation. BMJ Open. 2019 Nov 21;9(11):e025879. doi: 10.1136/bmjopen-2018-025879. PMID 31753865